CLINICAL TRIAL: NCT03406351
Title: Air Pollution, Asthma and Circadian Clocks
Acronym: APACC
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carsten Skarke, MD, Research Assistant Professor, University of Pennsylvania
Other Study IDs: IRB828728
Record Dates: First submitted 2018-01-14; First posted 2018-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Asthma; Healthy
MeSH Terms: conditions — Asthma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva, blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Asthma
  Interventions: Other: Observational
- Healthy: Matched controls
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational deep phenotyping physiological readouts

SUMMARY:
Societies become increasingly urban - more than half the world's population now lives in cities. Urbanization elevates anthropogenic (man-made) exposure to air pollutants. A clear association exists between exposure to air pollutants and exacerbations (worsening) of pre-existing asthma, incidence of nighttime asthma, difficulties with asthma control and increased disease risk. In 2012, the Public Health Management Corporation's Community Health Data Base estimated that 19.4% of adults in Philadelphia had asthma compared to a national prevalence of 7%.

Asthma has a clear temporal signal. A majority of asthma patients, up to 75%, reports nighttime awakenings due to worsened cough, wheeze and dyspnea. This time-of-day-dependent exacerbation of symptoms, coined nocturnal asthma, is associated with poorer disease control, more frequent medication, and higher asthma-related morbidity and mortality. Consequently, several pathophysiological mechanisms proposed for nocturnal asthma relate to circadian clock biology.

Lung function oscillates over the course of 24 hours, peaking around noon and reaching its nadir during early morning hours. Concentrations of air pollutants show oscillating patterns in urban settings.

In this clinical research study, the investigators start to address how spatiotemporal fluctuations in air pollutants relate to asthma. Mechanistically, the investigators wish to address the hypothesis that microRNAs (miRs) act as interface between asthma phenotypes, circadian clocks and environmental exposure.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age,
2. Physician's diagnosis of asthma,
3. Prescribed an inhaled-steroid-containing medication for asthma (ensuring the patient is believed to have at least moderate reversible airways obstruction by their physician),
4. severe persistent asthma according to the NHLBI Guidelines,
5. evidence of reversible airflow obstruction: (a) forced expiratory volume in 1 second (FEV1) <80% predicted at the time of or within 3 years of screening, and (b) improvement with bronchodilator: either (i) an increase of ≥15% and 200mL in FEV1 with asthma treatment over the previous 3 years or (ii) after 4 puffs of albuterol by MDI (or 2.5 mg by nebulizer), an increase in FEV1 or FVC ≥12% and 200 mL in FEV1 within 30 min at screening,
6. Own a smartphone.

Exclusion Criteria:

1. Severe psychiatric or cognitive problems (obvious mania, schizophrenia, significant mental retardation) making study conduct impossible. Formal psychiatric evaluations are outside of the scope; however, research coordinators will be trained to identify such cases followed by review of the PI. Patients can be referred to mental health facilities.
2. Past diagnosis of gastroesophageal reflux disease or obstructive sleep apnea,
3. Transmeridian travel across ≥2 time zones in the past month,
4. Planned transmeridian travel across more than ≥2 time zones during the planned study activities;
5. Use of oral or intravenous antibiotics in the past 6 months,
6. Episodes of bronchospasm in response to ultrasonic nebulizer treatment (to induce sputum collection non-invasively),
7. Any contraindication listed below in the separate paragraph "Contraindications for the use of CorTemp® Disposable Temperature Sensors";
8. Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
9. > 2 drinks of alcohol per day;
10. Use of illicit drugs;
11. Smoking;
12. Pregnant or nursing;
13. Avoid over-the-counter NSAID use 2 weeks prior to 48 hour session & during 48 hour session (Visit 3, Visit 4 & Visit 5);
14. Avoid Alcohol use 2 weeks prior to the 48 hour session and during the 3 day session (Visit 3, Visit 4 & Visit 5);
15. Vitamins use 1 week prior to and during the 48 hour session.
16. BMI > 30.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort 1: asthmatic patients (case); Cohort 2: matched healthy volunteers (control).
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Difference in expression levels of miR-142-3p in induced sputum from asthmatics versus controls | 48 hours
  Relative expression normalized to housekeeping genes (GAPDH, ACTB) plotted by Expression levels of miR-142-3p will be averaged from several measurements (morning, afternoon, evening, night with target times of 08:00, 14:00, 20:00, 02:00 +/- 1 hour) scheduled over 48 hours

SECONDARY OUTCOMES:
Concentration of ozone | 48 hours
  Concentrations of this air pollutant will be averaged in increments of one hour over the course of 48 hours
Concentration of the air pollutants CO, CO2, formaldehyde, particulate matter (PM) 1, PM2, PM10, tVOC (total volatile organic compounds) | 48 hours
  Concentrations of these air pollutants will be averaged in increments of one hour over the course of 48 hours
Disease expression of asthma measured how frequent asthma medication is used | 4 weeks
  The number of uses of asthma medication will determine severity of asthma
Circadian phase of cortisol | 48 hours
  Concentrations of cortisol in saliva will be determined in the morning, afternoon, evening, and night with target times of 08:00, 14:00, 20:00, 02:00 +/- 1 hour scheduled over 48 hours. Cosinor analysis will determine the circadian phase.

CONTACTS AND LOCATIONS:
Overall Officials: Garret FitzGerald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- See also: Researcher Carsten Skarke, MD — https://www.med.upenn.edu/apps/faculty/index.php/g275/p8152420